CLINICAL TRIAL: NCT01377610
Title: Long-acting Injectable Naltrexone Induction: A Randomized Trial of Outpatient Opioid Detoxification With Naltrexone vs. Buprenorphine
Brief Title: Improved Strategies for Outpatient Opioid Detoxification
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #6374/7250R; 2R01DA010746-09A1 (NIH)
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Opioid Dependence
Keywords: Outpatient detoxification; Opioid dependence; Naltrexone; Vivitrol; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; Buprenorphine; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Active Comparator): Standard 7-day buprenorphine induction and gradual taper from 8 mg to 0 mg followed on day 15 by Vivitrol injection
  Interventions: Drug: Buprenorphine; Drug: Vivitrol
- Oral naltrexone (Active Comparator): The naltrexone arm is a modification of our current inpatient naltrexone induction procedure, consisting of a single day of buprenorphine followed by a washout day and 4 days of ascending oral naltrexone doses. Followed on day 8 by Vivitrol injection.
  Interventions: Drug: oral naltrexone; Drug: Buprenorphine; Drug: Vivitrol

INTERVENTIONS:
Drug: oral naltrexone — Following detoxification with buprenorphine (one dy of 8 mg) followed by oral naltrexone (ascending taper to 25 mg), participants will receive Vivitrol injection on Day 8. Behavioral therapy sessions will be offered for five weeks.
  Other Names: buprenorphine and oral naltrexone followed by Vivitrol
  Arms: Oral naltrexone
Drug: Buprenorphine — Following detoxification with buprenorphine [8-mg buprenorphine (Day 1) tapering to 0 mg (Day 7)] participants will receive Vivitrol injection on Day 15. Behavioral therapy sessions will be offered for five weeks.
Drug: Vivitrol — dose of long-acting injectable naltrexone (Vivitrol 380 mg i.m. Injection)
  Other Names: long-acting injectable naltrexone

SUMMARY:
The investigators will randomize 210 opioid-dependent participants to one of two outpatient detoxification strategies: (1) a standard 7-day buprenorphine induction and gradual taper from 8 mg to 0 mg vs. (2) 7-day oral naltrexone induction; both groups will receive a single administration of a Vivitrol injection: at Day 8 for the naltrexone induction group and Day 15 for the buprenorphine group. The naltrexone arm is a modification of our current inpatient naltrexone induction procedure, consisting of a single day of buprenorphine followed by a washout day and 4 days of ascending oral naltrexone doses, prior to administering a dose of injectable naltrexone on Day 8. All participants will receive an intensive behavioral therapy for five weeks and will be followed for the subsequent 8 weeks to assess the longer-term outcome of the initial treatment. The primary outcome will be percentage of patients in each group successfully inducted onto Vivitrol. Key secondary outcomes will be 2-week abstinence at Weeks 4-5 (3rd and 4th weeks after Vivitrol injection), rates of completion of the 8-day detoxification, and percentage of patients in each group who return for additional Vivitrol injections in post-study follow-up. The main goal of this Stage 1a pilot study is to develop an improved outpatient opioid detoxification strategy, with particular relevance to newly diagnosed heroin addicts and prescription opioid abusers not seeking long-term agonist maintenance.

Specific Aim #1: To develop procedures for outpatient opioid detoxification which include naltrexone to facilitate detoxification.

Specific Aim #2: To compare injectable naltrexone induction rates between the naltrexone and buprenorphine groups following short-term outpatient opioid detoxification approach for initiating treatment for opioid dependence.

DETAILED DESCRIPTION:
We are proposing a randomized, parallel-groups 5-week study of relapse prevention in detoxified opioid-dependent individuals. This trial represents an initial test of the feasibility and efficacy of an outpatient opioid detoxification strategy employing induction onto long-acting naltrexone (Vivitrol), in combination with the recently adapted version of Behavioral Naltrexone Therapy for Depot Naltrexone (Depot-BNT). Participants will be randomized into one of two outpatient detoxification strategies: (1) standard 7-day buprenorphine induction and taper from 8 mg to 0 mg (N=33), followed on Day 15 by a naloxone challenge and a dose of long-acting injectable naltrexone (Vivitrol) (consistent with the FDA-approved recommendation of 7 or more days between last opioid dose and Vivitrol induction) vs. (2) a modification of our current inpatient naltrexone induction procedure, consisting of a single day of buprenorphine followed by a washout day and 4 days of ascending oral naltrexone doses, followed by long-acting injectable naltrexone (Vivitrol) 380 mg on Day 8 (N=67). We are seeking to obtain Vivitrol samples from Alkermes; if we are successful in obtaining such samples, we will offer all participants who complete the study a second injection 4 weeks after the first, and a third injection will be offered at Week 12. All participants will receive an intensive behavioral therapy for five weeks and will be followed for up to 24 weeks to assess the long-term outcome of the initial treatment. Study assessments will be collected at baseline and at each study visit (twice weekly in Weeks 2-5; weekly in Weeks 6-9 for participants who receive a second Vivitrol injection and participate in follow-up care). Repeated assessments will also be completed at one and four months following the end of treatment. The primary aim of this study is to test the hypothesis that an outpatient opioid detoxification strategy using naltrexone will increase the likelihood of successful induction onto long-acting injectable naltrexone, compared to a buprenorphine taper in opioid-dependent patients. The primary outcome measure will be percentage in each treatment group (oral naltrexone vs. buprenorphine taper) receiving the Vivitrol injection at Day 8 or 15. Key secondary outcomes will be: two-week opioid abstinence during Weeks 4-5, retention in the 8-day detoxification procedure (time to dropout) and severity of opiate withdrawal during the first 5 weeks of treatment. We anticipate that the outpatient opioid detoxification method developed in this project will be uniquely suited to the needs of the rapidly expanding population of prescription opioid-abusing individuals seeking an alternative to opioid agonist maintenance. The current proposal will also yield important data on how to improve long-term outcomes for the buprenorphine taper method of opioid detoxification, through the addition of long-acting naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current opiate dependence disorder of at least six months duration, supported by urine toxicology OR COWS score > or =6 OR Naloxone Challenge .
* Seeking treatment for opioid dependence.
* In otherwise good health based on complete medical history and physical examination
* Able to give written informed consent.

Exclusion Criteria:

* Methadone maintenance treatment or regular use of illicit methadone (> 30 mg per week).
* Maintenance on, or regular use of buprenorphine or other long-acting narcotic agonists
* Active medical illness which might make participation hazardous, such as untreated hypertension, acute hepatitis with AST or ALT > 3 times normal, AIDS, unstable diabetes.
* Severe psychiatric illness (psychotic disorder, major depression, suicide risk or 1 or more suicide attempts within the past year.)
* Physiologically dependent on alcohol or sedative-hypnotics
* History of allergic or adverse reaction to buprenorphine, naltrexone, naloxone, clonidine, or clonazepam.
* Chronic pain requiring opioid analgesia or anticipated surgery necessitating opioid medications
* AIDS dementia or other chronic organic mental disorder
* Pregnancy, lactation, failure to use contraception
* History of accidental drug overdose in the last 3 years as defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2011-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in each group successfully inducted onto Vivitrol | Completion of 7-day detoxification
  Comparison of the percentage of patients assigned to each detoxification group (oral naltrexone vs. buprenorphine) who receive Vivitrol at the completion of detoxification.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, M.D., Principal Investigator — Columbia University and NYSPI
Locations (1):
- Substance Treatment and Research Service (STARS), Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Sullivan M, Bisaga A, Pavlicova M, Choi CJ, Mishlen K, Carpenter KM, Levin FR, Dakwar E, Mariani JJ, Nunes EV. Long-Acting Injectable Naltrexone Induction: A Randomized Trial of Outpatient Opioid Detoxification With Naltrexone Versus Buprenorphine. Am J Psychiatry. 2017 May 1;174(5):459-467. doi: 10.1176/appi.ajp.2016.16050548. Epub 2017 Jan 10. PMID 28068780
- See also: stars website — http://stars.columbia.edu